CLINICAL TRIAL: NCT07242781
Title: A Phase 1, Open-label, 2-part, Fixed-sequence, Crossover Study to Evaluate the Effect of Cytochrome P450 (CYP) 3A Inhibitor (Itraconazole) and Inducer (Rifampin) on the Pharmacokinetics of AR-LDD (BMS-986365) in Healthy Adult Male Participants
Brief Title: A Study to Evaluate the Effect of Itraconazole and Rifampin on the Drug Levels of AR-LDD (BMS-986365) in Healthy Adult Male Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CA071-1006
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers
Keywords: Healthy male volunteers; BMS-986365; CC-94676; Itraconazole; Rifampin; Pharmacokinetics; Crossover; Open-label
MeSH Terms: interventions — Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A (Safety Lead-in Group) (Experimental)
  Interventions: Drug: BMS-986365; Drug: Itraconazole
- Part A, Period 1 (Experimental)
  Interventions: Drug: BMS-986365
- Part A, Period 2 (Experimental)
  Interventions: Drug: BMS-986365; Drug: Itraconazole
- Part B, Period 1 (Experimental)
  Interventions: Drug: BMS-986365
- Part B, Period 2 (Experimental)
  Interventions: Drug: BMS-986365; Drug: Rifampin

INTERVENTIONS:
Drug: BMS-986365 — Specified dose on specified days
  Other Names: AR-LDD, CC-94676
Drug: Itraconazole — Specified dose on specified days
  Other Names: SPORANOX®
  Arms: Part A (Safety Lead-in Group); Part A, Period 2
Drug: Rifampin — Specified dose on specified days
  Arms: Part B, Period 2

SUMMARY:
The purpose of this study is to evaluate the effect of Itraconazole and Rifampin on the drug levels of AR-LDD (BMS-986365) in healthy adult male participants.

ELIGIBILITY:
Inclusion Criteria

* Participants must be male, at the time of signing the Informed Consent Form (ICF), have a Body Mass Index (BMI) of 18.0 to 32.0 kg/m2; and healthy as determined by medical history, PE, vital signs, 12-lead ECG, transthoracic echocardiogram (TTE) and clinical laboratory assessments.

Exclusion Criteria

* Participants must not have any significant or chronic illness.
* Participants must not have a prior history of heart failure, ischemic heart diseases, serious cardiac arrythmias, or prolonged QT interval.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-06-14 (Estimated); Study Completion 2026-06-14 (Estimated)

PRIMARY OUTCOMES:
Part A: Maximum Observed Plasma Concentration (Cmax) of BMS-986365 | Up to approximately Day 32
Part A: Cmax of BMS-986365 Without Itraconazole | Up to approximately Day 32
Part A: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC(0-T)) of BMS-986365 With Itraconazole | Up to approximately Day 32
Part A: AUC(0-T) of BMS-986365 Without Itraconazole | Up to approximately Day 32
Part A: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinite Time (AUC(INF)) of BMS-986365 | Up to approximately Day 32
Part A: AUC(INF) of BMS-986365 Without Itraconazole | Up to approximately Day 32
Part B: Cmax of BMS-986365 With Rifampin | Up to approximately Day 37
Part B: Cmax of BMS-986365 Without Rifampin | Up to approximately Day 37
Part B: AUC(INF) of BMS-986365 With Rifampin | Up to approximately Day 37
Part B: AUC(INF) of BMS-986365 Without Rifampin | Up to approximately Day 37
Part B: AUC(0-T) of BMS-986365 With Rifampin | Up to approximately Day 37
Part B: AUC(0-T) of BMS-986365 Without Rifampin | Up to approximately Day 37

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to approximately Day 89
Number of Participants With Serious Adverse Events (SAEs) | Up to approximately Day 89
Number of Participants With AEs Leading to Drug/Study Discontinuation | Up to approximately Day 89
Number of Participants With Clinically Significant Vital Sign Measurements | Up to approximately Day 77
Number of Participants With Clinically Significant Laboratory Safety Tests | Up to approximately Day 77
  Laboratory safety tests include hematology, chemistry, and urinalysis.
Number of Participants With Clinically Significant 12-lead Electrocardiogram (ECG) Abnormalities | Up to approximately Day 77
Number of Participants With Clinically Significant Physical Examination (PE) Abnormalities | Up to approximately Day 77
Change From Baseline of Corrected QT Interval (QTc) Post Dose of BMS-986365 | Up to approximately Day 77
Part A: Change From Baseline of QTc Post Dose of BMS-986365 With Itaconazole | Up to approximately Day 72
Part B: Change From Baseline of QTc Post Dose of BMS-986365 With Rifampin | Up to approximately Day 77
Time of Maximum Observed Plasma Concentration (Tmax) of BMS-986365 | Up to approximately Day 77
Apparent Terminal Plasma Half-life (T-HALF) of BMS-986365 | Up to approximately Day 77
Apparent Total Body Clearance (CLT/F) of BMS-986365 | Up to approximately Day 77
Apparent Volume of Distribution of Terminal Phase (Vz/F) of BMS-986365 | Up to approximately Day 77

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Syneos Health Clinic, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html